CLINICAL TRIAL: NCT03070730
Title: A Double-Blinded, Placebo-Controlled Study To Assess Hemodynamic Changes, Orthostatic Tolerance, Out-Patient Fatigue And Quality Of Life In Neuropathic And Non-Neuropathic POTS Patients In Response To Adrenoreceptor Agonist And Antagonist
Brief Title: Hemodynamic Response of Neuropathic And Non-Neuropathic POTS Patients To Adrenoreceptor Agonist And Antagonist
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment was slow and subjects declined participation after signing the ICF.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Roy Freeman, MD, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011P000246; R01HL059459 (NIH)
Record Dates: First submitted 2012-02-27; First posted 2017-03-06 (Actual); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance
Keywords: Tachycardia; orthostatic symptoms; autonomic reflex
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance; Tachycardia | interventions — Droxidopa; Atenolol

STUDY DESIGN:
Intervention Model Description: The study design is a "double-dummy" design. While during two of the three trial arms the patients take an active study drug and a placebo, there is also an arm where patients take only placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atenolol (Other): In this arm subjects are randomized to atenolol 50 mg qd, droxidopa 100 mg/300 mg tid and placebo tid.
  Atenolol is used to examine the effect of non-selective beta adrenoreceptor antagonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia patients.
  Droxidopa is used to examine the effect of direct alpha-1 adrenoreceptor agonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia (POTS) patients.
  Interventions: Drug: Droxidopa; Drug: Atenolol; Drug: Placebos
- Placebos (Other): In this arm subjects are randomized to placebo tid.
  Placebo is used to control the administration effect.
  Interventions: Drug: Placebos
- Droxidopa (Other): In this arm subjects are randomized to droxidopa 100 mg/300 mg tid, atenolol 50 mg qd, and placebo tid.
  Atenolol is used to examine the effect of non-selective beta adrenoreceptor antagonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia patients.
  Droxidopa is used to examine the effect of direct alpha-1 adrenoreceptor agonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia (POTS) patients.
  Interventions: Drug: Droxidopa; Drug: Atenolol; Drug: Placebos

INTERVENTIONS:
Drug: Droxidopa — Droxidopa: 100 mg or 300 mg t.i.d
  Other Names: Northera
  Arms: Atenolol; Droxidopa
Drug: Atenolol — Atenolol: 50 mg Q.D.
  Other Names: Tenormin
  Arms: Atenolol; Droxidopa
Drug: Placebos — Placebo: t.i.d
  Other Names: placebo

SUMMARY:
The purpose of this study is to test the hypothesis that patients with non-neuropathic POTS will have different responsiveness than patients with neuropathic POTS to direct alpha-1 adrenoreceptor agonist therapy (droxidopa) and to non-selective beta-adrenoreceptor antagonist therapy (atenolol).

The specific goal of this protocol is to investigate the effect of atenolol and droxidopa on cardiovascular autonomic functions such as cardiovagal control, sympathetic nerve activity, and sympathetic vascular transduction, systemic hemodynamic response to orthostatic stress and on the quality of life in neuropathic and non-neuropathic patients with postural tachycardia syndrome (POTS).

Standardized tests are used to assess cardiovagal control function, sympathetic nerve activity, sympathetic vascular transduction, systemic hemodynamic response to head-up tilt test and standardized questionnaires to assess the quality of life in patients with POTS.

The cardiovagal, sympathetic and hemodynamic measurements are performed after and during drug administration. To control the effect of medications placebo is used on separate testing visits. The order of drugs and placebo is randomized.

DETAILED DESCRIPTION:
The pathophysiological basis of postural tachycardia syndrome (POTS) is not well elucidated. The most widely recognized primary cause of POTS is a "restricted" or "selective" peripheral neuropathy - neuropathic POTS. Several lines of evidence point to a restricted peripheral neuropathy, specifically sympathetic denervation in the lower hemibody, as a cause of POTS. These include venous denervation, impaired distal sudomotor dysfunction, lower norepinephrine spillover in the legs than the arms. However, not all POTS patients have peripheral neuropathy. Proposed pathogenic etiologies for non-neuropathic POTS include deconditioning, low-grade inflammation and oxidative stress. Neuropathic POTS is present in 33% of patients while non-neuropathic POTS is present in 67% of patients.

The most frequent neuropathic feature in the neuropathic POTS group is decreased sweat output measured by quantitative sudomotor axon reflex test. Headache and gastrointestinal symptoms (such as abdominal pain, bloating, nausea and constipation) are also more prevalent in the neuropathic than in the non-neuropathic POTS group, suggesting more global differences between the two populations.

In relation to the ambiguous pathophysiological basis, there is no definitive treatment for POTS. There are reports of improvements in hemodynamic measures and symptoms of orthostatic tolerance with pharmacologic agents that include intravenous saline, intravenous phenylephrine, midodrine, octreotide, erythropoietin, pyridostigmine, and betablockade. The therapy is however frequently disappointing. Furthermore, there are no reported long-term studies of medications to treat POTS and there are no reports of the effects of any intervention on fatigue or quality of life.

The most widely used agents to treat POTS, the alpha-adrenoreceptor agonist midodrine, and the beta blockers, paradoxically have agonistic and antagonistic effects on the autonomic nervous system. Responses to these drugs are inconsistent and there are no delineated predictors of the response in POTS patients.

The comparison of therapeutic interventions in this protocol are based on the rationale that while alpha-adrenoreceptor agonists are thought to be more effective in neuropathic POTS - a disorder characterized by a compensatory increase in sympathetic outflow in which sympatholysis may be counterproductive, beta-adrenoreceptor antagonists are thought to be more effective in non-neuropathic POTS - a disorder that could be characterized by increased central sympathetic outflow due to impaired sympathetic inhibition.

This protocol uses droxidopa, which is converted to direct adrenoreceptor agonist, norepinephrine. The protocol also uses beta-adrenoreceptor antagonist, the non-selective atenolol.

This is a randomized, double-blind, placebo-controlled, cross-over experimental study with three trial arms, according to the two medications (droxidopa and atenolol) and the placebo. The trial is performed in the Center for Autonomic and Peripheral Nerve Disorders at the Beth Israel Deaconess Medical Center.

The study consists of 10 visits:

* screening visit,
* testing days to define drug sensitivity
* classification day
* autonomic testing visits
* follow-up visits

Screening visit (Visit 1) includes

* Consenting procedure
* Review of medical history
* Review of all current medications, prescription and over the counter
* Physical and neurological examinations
* Measure height, weight, temperature and vital signs
* 12-lead ECG
* Baseline autonomic tests
* Blood labs
* Serum pregnancy testing for women of childbearing potential
* Patients are able to take PO medications

Drug Sensitivity Visit (Visit 2 and 3) On the first visit, patients receive one 100 mg droxidopa while on the second visit patients receive one 300 mg test dose of droxidopa to define their response to the drug. The drug administration is preceded and followed by heart rate and blood pressure measurements and side effect monitoring. The two consecutive visits are made within a period of 3 days. The goal of sensitivity visit is to determine if a patient has any sign of denervation supersensitivity in response to droxidopa. The patient is considered to have denervation supersensitivity if systolic blood pressure is greater than 180 mmHg or diastolic blood pressure is greater than 110 mmHg after 3 minutes of standing or after 5 minutes of sitting or the patient is unable to tolerate the side effects believed to be related to the drug.

Patient classification visit (Visit 4) includes

* Quantitative Direct and Indirect testing of Sudomotor Function (QDIRT)
* Quantitative Sudomotor Axon Reflex Testing (QSART)
* Quantitative Sensory Testing (QST)
* Punch skin biopsy
* Questionnaires (Chronic Fatigue Screening Form, Fatigue Severity Scale, Chalder Fatigue Questionnaire, etc., see Questionnaires section)

Autonomic Evaluation Visits (Visit 5, 7 and 9) include

* Urine pregnancy test for women of child-bearing potential
* Setup and instrumentation
* Blood draw for hormones and catecholamines (Visit 5 only)
* Microneurography procedure
* Drug/placebo administration
* Deep breathing test
* Paced breathing test
* Modified Oxford test
* Sympathetic transduction
* Static exercise
* Tilt table test

Primary outcome measure of autonomic evaluation visit is maximum postural tachycardia while secondary outcome measure of autonomic evaluation visit are blood pressure, heart rate, vascular resistance, muscle sympathetic nerve activity.

Follow-up testing visits (Visit 6, 8 and 10) include

* Medical history
* Physical examination
* Vital signs
* EKG
* Blood pressure measurement
* Tilt table test

Primary outcome measure of follow-up testing visits is the fatigue score on the Chalder Fatigue questionnaire while secondary outcome measures of follow-up testing visits are the scores on the physical functioning subscale of the SF-36 questionnaire, 7 item patient global impression of change, the Hospital Anxiety and Depression Scales, the Checklist Individual Strength (CIS), Multidimensional Fatigue Inventory (MFI), the Fatigue Severity Scale, the EuroQOL, the HADS and anxiety scores. The Orthostatic Intolerance Questionnaire - a unique validated questionnaire is used to assess orthostatic intolerance symptoms and quality of life-related to orthostatic intolerance.

ELIGIBILITY:
Inclusion Criteria:

* CDC criteria for chronic fatigue syndrome
* Evidence of postural tachycardia syndrome with symptoms of orthostatic intolerance

Exclusion Criteria:

* Pregnant or lactating females. The administration of droxidopa is harmful to the fetus
* Concomitant therapy with anticholinergic, alpha-, and beta-adrenergic antagonists or other medications that affect autonomic function
* Clinically significant coronary artery, cerebrovascular or peripheral vascular disease
* Cardiac arrhythmias
* Systemic illness that might affect autonomic function such as congestive heart failure, hypertension, renal, pulmonary, and hepatic disease, anemia, malignancies, thyroid disease, and alcoholism
* Severe depression, severe anxiety disorder (score of on the Beck Depression Inventory > 29 or score on the Beck Anxiety Inventory of ≥ 36) or psychosis
* Antidepressant treatment by MAO inhibitors within 2 weeks before the study
* Glaucoma
* Liver disease
* Subjects with a history of reaction to local anesthetic will be excluded from the study
* Subjects who have a history of any bleeding disorders or significantly impaired wound healing will be excluded. Subjects who are using any medications such as Coumadin or Plavix will be also excluded
* Subjects who are currently enrolled in any other studies using investigational products

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2012-12-18 (Actual); Study Completion 2014-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Freeman, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Center for Autonomic and Peripheral Nerve Disorders - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
NIH Grant Policy on Sharing of Unique Research Resources including the Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources.

REFERENCES:
- [Background] Jacob G, Biaggioni I. Idiopathic orthostatic intolerance and postural tachycardia syndromes. Am J Med Sci. 1999 Feb;317(2):88-101. doi: 10.1097/00000441-199902000-00003. PMID 10037112
- [Background] Karas B, Grubb BP, Boehm K, Kip K. The postural orthostatic tachycardia syndrome: a potentially treatable cause of chronic fatigue, exercise intolerance, and cognitive impairment in adolescents. Pacing Clin Electrophysiol. 2000 Mar;23(3):344-51. doi: 10.1111/j.1540-8159.2000.tb06760.x. PMID 10750135
- [Background] Stewart JM. Autonomic nervous system dysfunction in adolescents with postural orthostatic tachycardia syndrome and chronic fatigue syndrome is characterized by attenuated vagal baroreflex and potentiated sympathetic vasomotion. Pediatr Res. 2000 Aug;48(2):218-26. doi: 10.1203/00006450-200008000-00016. PMID 10926298
- [Background] Schondorf R, Low PA. Idiopathic postural orthostatic tachycardia syndrome: an attenuated form of acute pandysautonomia? Neurology. 1993 Jan;43(1):132-7. doi: 10.1212/wnl.43.1_part_1.132. PMID 8423877
- [Background] Jacob G, Costa F, Shannon JR, Robertson RM, Wathen M, Stein M, Biaggioni I, Ertl A, Black B, Robertson D. The neuropathic postural tachycardia syndrome. N Engl J Med. 2000 Oct 5;343(14):1008-14. doi: 10.1056/NEJM200010053431404. PMID 11018167
- [Background] Streeten DH. Pathogenesis of hyperadrenergic orthostatic hypotension. Evidence of disordered venous innervation exclusively in the lower limbs. J Clin Invest. 1990 Nov;86(5):1582-8. doi: 10.1172/JCI114878. PMID 2243132
- [Background] Low PA, Novak V, Spies JM, Novak P, Petty GW. Cerebrovascular regulation in the postural orthostatic tachycardia syndrome (POTS). Am J Med Sci. 1999 Feb;317(2):124-33. doi: 10.1097/00000441-199902000-00007. PMID 10037116
- [Background] Freeman R, Lirofonis V, Farquhar WB, Risk M. Limb venous compliance in patients with idiopathic orthostatic intolerance and postural tachycardia. J Appl Physiol (1985). 2002 Aug;93(2):636-44. doi: 10.1152/japplphysiol.00817.2001. PMID 12133874
- [Background] Shannon JR, Flattem NL, Jordan J, Jacob G, Black BK, Biaggioni I, Blakely RD, Robertson D. Orthostatic intolerance and tachycardia associated with norepinephrine-transporter deficiency. N Engl J Med. 2000 Feb 24;342(8):541-9. doi: 10.1056/NEJM200002243420803. PMID 10684912
- [Background] Al-Shekhlee A, Lindenberg JR, Hachwi RN, Chelimsky TC. The value of autonomic testing in postural tachycardia syndrome. Clin Auton Res. 2005 Jun;15(3):219-22. doi: 10.1007/s10286-005-0282-7. PMID 15944872
- [Background] Stewart JM, Munoz J, Weldon A. Clinical and physiological effects of an acute alpha-1 adrenergic agonist and a beta-1 adrenergic antagonist in chronic orthostatic intolerance. Circulation. 2002 Dec 3;106(23):2946-54. doi: 10.1161/01.cir.0000040999.00692.f3. PMID 12460877
- [Background] Gordon VM, Opfer-Gehrking TL, Novak V, Low PA. Hemodynamic and symptomatic effects of acute interventions on tilt in patients with postural tachycardia syndrome. Clin Auton Res. 2000 Feb;10(1):29-33. doi: 10.1007/BF02291387. PMID 10750641
- [Background] Freitas J, Santos R, Azevedo E, Costa O, Carvalho M, de Freitas AF. Clinical improvement in patients with orthostatic intolerance after treatment with bisoprolol and fludrocortisone. Clin Auton Res. 2000 Oct;10(5):293-9. doi: 10.1007/BF02281112. PMID 11198485
- [Background] Gibbons CH, Vernino SA, Kaufmann H, Freeman R. L-DOPS therapy for refractory orthostatic hypotension in autoimmune autonomic neuropathy. Neurology. 2005 Oct 11;65(7):1104-6. doi: 10.1212/01.wnl.0000178980.83477.14. PMID 16217067
- [Background] Low PA, Opfer-Gehrking TL, Textor SC, Benarroch EE, Shen WK, Schondorf R, Suarez GA, Rummans TA. Postural tachycardia syndrome (POTS). Neurology. 1995 Apr;45(4 Suppl 5):S19-25. PMID 7746369
- [Background] Grubb BP, Kosinski DJ, Boehm K, Kip K. The postural orthostatic tachycardia syndrome: a neurocardiogenic variant identified during head-up tilt table testing. Pacing Clin Electrophysiol. 1997 Sep;20(9 Pt 1):2205-12. doi: 10.1111/j.1540-8159.1997.tb04238.x. PMID 9309745
- [Background] Sandroni P, Opfer-Gehrking TL, McPhee BR, Low PA. Postural tachycardia syndrome: clinical features and follow-up study. Mayo Clin Proc. 1999 Nov;74(11):1106-10. doi: 10.4065/74.11.1106. PMID 10560597
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Paffenbarger RS Jr, Blair SN, Lee IM, Hyde RT. Measurement of physical activity to assess health effects in free-living populations. Med Sci Sports Exerc. 1993 Jan;25(1):60-70. doi: 10.1249/00005768-199301000-00010. PMID 8423758
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Moss-Morris R, Sharon C, Tobin R, Baldi JC. A randomized controlled graded exercise trial for chronic fatigue syndrome: outcomes and mechanisms of change. J Health Psychol. 2005 Mar;10(2):245-59. doi: 10.1177/1359105305049774. PMID 15723894

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants that were enrolled in the study were excluded from the study because they either did not meet eligibility criteria or decided not to participate.
Groups:
- Atenolol: In this arm subjects are randomized to atenolol 50 mg qd, droxidopa 100 mg/300 mg tid and placebo tid.
  Atenolol is used to examine the effect of non-selective beta adrenoreceptor antagonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia patients.
  Droxidopa is used to examine the effect of direct alpha-1 adrenoreceptor agonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia (POTS) patients.
  Droxidopa: Droxidopa: 100 mg or 300 mg t.i.d
  Atenolol: Atenolol: 50 mg Q.D.
  Placebos: Placebo: t.i.d
- Placebos: In this arm subjects are randomized to placebo tid.
  Placebo is used to control the administration effect.
  Placebos: Placebo: t.i.d
- Droxidopa: In this arm subjects are randomized to droxidopa 100 mg/300 mg tid, atenolol 50 mg qd, and placebo tid.
  Atenolol is used to examine the effect of non-selective beta adrenoreceptor antagonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia patients.
  Droxidopa is used to examine the effect of direct alpha-1 adrenoreceptor agonist on primary and secondary endpoints in neuropathic and non-neuropathic postural tachycardia (POTS) patients.
  Droxidopa: Droxidopa: 100 mg or 300 mg t.i.d
  Atenolol: Atenolol: 50 mg Q.D.
  Placebos: Placebo: t.i.d
Period: Overall Study
Arm/Group | Atenolol | Placebos | Droxidopa
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants that were enrolled in the study were not randomized. They did not meet eligibility criteria, or decided not to participate.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atenolol | Placebos | Droxidopa | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Customized | 0 | 0 | 0 |
Sex: Female, Male
  Female | 0 | 0 | 0 |
  Male | 0 | 0 | 0 |
Race (NIH/OMB)
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal Postural Tachycardia During Tilt
Description: Maximal postural tachycardia is the maximum heart rate during a 20-min tilt table test.
Time Frame: Up to 3 days after randomization
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

2. Primary Outcome: Change Maximal Postural Tachycardia During Tilt
Description: Maximal postural tachycardia is the maximum heart rate during a 20-min tilt table test.
Time Frame: 2 weeks after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

3. Primary Outcome: Change Maximal Postural Tachycardia During Tilt
Description: Maximal postural tachycardia is the maximum heart rate during a 20-min tilt table test.
Time Frame: 2 weeks after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

4. Primary Outcome: Change in Fatigue Score on the Chalder Fatigue Questionnaire From Baseline
Description: A 14 item self-report questionnaire. Subjects respond on a continuum of 1 to 4 questions evaluating fatigue intensity while distinguishing physical from mental fatigue.
Time Frame: up to 3 days after randomization
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

5. Primary Outcome: Change in Fatigue Score on the Chalder Fatigue Questionnaire From Baseline
Description: as for outcome 4
Time Frame: 2 weeks after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

6. Primary Outcome: Change in Fatigue Score on the Chalder Fatigue Questionnaire From Baseline
Description: as for outcome 4
Time Frame: 2 weeks after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

7. Secondary Outcome: Change in Blood Pressure From Baseline
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

8. Secondary Outcome: Change in Blood Pressure From Baseline
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

9. Secondary Outcome: Change in Blood Pressure From Baseline
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

10. Secondary Outcome: Change in Heart Rate From Baseline
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

11. Secondary Outcome: Change in Heart Rate From Baseline
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

12. Secondary Outcome: Change in Heart Rate From Baseline
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

13. Secondary Outcome: Change in Vascular Resistance From Baseline
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

14. Secondary Outcome: Change in Vascular Resistance From Baseline
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

15. Secondary Outcome: Change in Vascular Resistance From Baseline
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

16. Secondary Outcome: Change in Muscle Sympathetic Nerve Activity From Baseline
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

17. Secondary Outcome: Change in Muscle Sympathetic Nerve Activity From Baseline
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

18. Secondary Outcome: Change in Muscle Sympathetic Nerve Activity From Baseline
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

19. Secondary Outcome: Change in Physical Functioning-SF-36 Q From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the SF-36 questionnaire.
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

20. Secondary Outcome: Change in Physical Functioning-SF-36 Q From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the SF-36 questionnaire.
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

21. Secondary Outcome: Change in Physical Functioning-SF-36 Q From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the SF-36 questionnaire.
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

22. Secondary Outcome: Change in Physical Functioning- 7 Item Patient Global Impression of Change From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the 7 item patient global impression of change with items anchored by :very much better" to "very much worse".
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

23. Secondary Outcome: Change in Physical Functioning- 7 Item Patient Global Impression of Change From Baseline
Description: as for outcome 22
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

24. Secondary Outcome: Change in Physical Functioning- 7 Item Patient Global Impression of Change From Baseline
Description: as for outcome 22
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

25. Secondary Outcome: Change in Physical Functioning- HADS From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the Hospital Anxiety and Depression Scales.
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

26. Secondary Outcome: Change in Physical Functioning- HADS From Baseline
Description: as for outcome 25
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

27. Secondary Outcome: Change in Physical Functioning- HADS From Baseline
Description: as for outcome 25
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

28. Secondary Outcome: Change in Physical Functioning-CIS From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the Checklist Individual Strength (CIS).
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

29. Secondary Outcome: Change in Physical Functioning-CIS From Baseline
Description: as for outcome 28
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

30. Secondary Outcome: Change in Physical Functioning-CIS From Baseline
Description: as for outcome 28
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

31. Secondary Outcome: Change in Physical Functioning-MFI From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the Multidimensional Fatigue Inventory (MFI).
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

32. Secondary Outcome: Change in Physical Functioning-MFI From Baseline
Description: as for outcome 31
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

33. Secondary Outcome: Change in Physical Functioning-MFI From Baseline
Description: as for outcome 31
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

34. Secondary Outcome: Change in Physical Functioning-FSS From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the Fatigue Severity Scale.
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

35. Secondary Outcome: Change in Physical Functioning-FSS From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the Fatigue Severity Scale.
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

36. Secondary Outcome: Change in Physical Functioning-FSS From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the Fatigue Severity Scale.
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

37. Secondary Outcome: Change in Physical Functioning-EuroQOL From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the EuroQOL.
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

38. Secondary Outcome: Change in Physical Functioning-EuroQOL From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the EuroQOL.
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

39. Secondary Outcome: Change in Physical Functioning-EuroQOL From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the EuroQOL.
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

40. Secondary Outcome: Change in Physical Functioning-OI From Baseline
Description: Measures of follow up testing will be the scores on the physical functioning subscale of the Orthostatic Intolerance Questionnaire.
Time Frame: 1 week after first intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

41. Secondary Outcome: Change in Physical Functioning-OI From Baseline
Description: as for outcome 40
Time Frame: 1 week after second intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

42. Secondary Outcome: Change in Physical Functioning-OI From Baseline
Description: as for outcome 40
Time Frame: 1 week after third intervention
Arm/Group | Atenolol | Placebos | Droxidopa
Number analyzed (Participants) | 0 | 0 | 0
Value | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Atenolol | Placebos | Droxidopa
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The trial was terminated early due to difficulties in the recruitment process. Subjects were found to be ineligible, or decided not to participate in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No